CLINICAL TRIAL: NCT06157073
Title: A Randomized, Controlled Trial to Evaluate the Efficacy and Safety of Fully Automated Closed-loop Ventilator Versus Conventional Open-loop Ventilator in Ventilated Patients in the Emergency Department
Brief Title: Efficacy and Safety of Automated Closed-loop Ventilator vs Conventional Open-loop Ventilator in the Emergency Department
Acronym: AVAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Khadijah Poh Yuen Yoong, Consultant Emergency Physician, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023317-12254; NMRR ID-23-03290-LRC (Registry Identifier: National Medical Research Register)
Record Dates: First submitted 2023-11-16; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Ventilator Lung; Mechanical Ventilation Complication; Ventilator-Induced Lung Injury; ARDS
Keywords: mechanical ventilation; closed loop ventilator; open loop ventilator; emergency department
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Emergencies

STUDY DESIGN:
Intervention Model Description: Subjects who meet all criteria for enrolment will be randomized in a 1:1 allocation ratio to receive either open-loop ventilator (OLV) or closed-loop ventilator (CLV). Randomization will be stratified by the respiratory pathology present: normal lung, hypercapnic respiratory failure and decreased lung compliance. Randomization sequence will be generated using a web-based randomisation software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open-loop ventilator (Active Comparator): Prior to the rapid sequence intubation, patients' gender and height are set on the ventilator. The physician in-charge will setup the ventilator based on the lung condition, following the research protocol. Patients will be connected to this ventilator upon securing the airway. Ventilator setting parameters will be manually adjusted by the in-charge physician following local guidelines.
  Interventions: Device: Open-loop ventilator
- Closed-loop ventilator (Experimental): Prior to the rapid sequence intubation, patients' gender and height are set on the ventilator. Patients' condition settings are selected depending on the lung condition. The sensors for end-tidal carbon dioxide (EtCO2) and oxygen saturation (SpO2) will be connected. Patients will be connected to this ventilator upon securing the airway. Ventilator setting parameters will be set following the study protocol.
  Interventions: Device: Closed-loop ventilator

INTERVENTIONS:
Device: Closed-loop ventilator — Fully automated closed-loop ventilator using the INTELLIVENT software
  Arms: Closed-loop ventilator
Device: Open-loop ventilator — Conventional closed-loop ventilator with manual adjustments by the physician in charge
  Arms: Open-loop ventilator

SUMMARY:
Patients presenting to the emergency department (ED) may require breathing support with machines depending on the condition. Throughout the breathing support, the settings on the breathing machines will be tailored to the patient's requirements. These settings are manually adjusted by trained physicians. Currently, there are machines which can automatically change the settings based on real-time specific information obtained from the patient. This study aims to compare the use of machines which require manual adjustments (open-loop conventional ventilators) and machines which can automatically change the settings (closed-loop automated ventilators). Patients will be carefully selected to ensure no harm is caused whilst delivering the best care. This study will look into the duration when patients are receiving optimum settings and levels of oxygen and carbon dioxide in the blood. The outcomes of this study would allow us to identify methods to improve patient care.

DETAILED DESCRIPTION:
Invasive mechanical ventilation is a lifesaving intervention for patients with respiratory failure in the emergency department (ED). Recent technological advancements have introduced closed-loop automated ventilators as a potential alternative to open-loop conventional ventilators. However, the efficacy and safety of closed-loop automated ventilators in the emergency setting remains understudied. This research aims to evaluate the efficacy and safety of closed-loop automated ventilator compared to open-loop conventional ventilator in intubated and ventilated patients in the ED.

A randomized controlled trial will be conducted in an ED of a tertiary university-affiliated hospital. Eligible patients are 18 years or older, decision made by treating physicians to intubate and mechanically ventilate. Some of exclusion criteria are pregnancy, heart failure, metabolic acidosis, circulatory shock, life-threatening asthma and morbid obesity. The primary measure of efficacy is the duration of ventilation within a predefined range of acceptable respiratory parameters between automated and conventional ventilation. Secondary outcome measures are; number of manual adjustments required to attain targeted settings in automated and conventional ventilators, PaO2/FiO2 ratio (PF ratio), arterial blood gas results, vital signs, breath-by-breath analysis, and rate of ventilator dyssynchrony. The ventilator used in the intervention arm is the closed-loop automated ventilator Hamilton C6s INTELLIVENT-ASV (Hamilton Medical AG, Switzerland). Hamilton C1 ASV is chosen as the open-loop conventional comparator as it is similar to Hamilton C6s INTELLIVENT-ASV, without the INTELLIVENT software.

Based on Lellouche et al, the calculated total sample size with a dropout rate of 10% is 132. The data is analysed based on the intention-to-treat (ITT) and per-protocol (PP) principles. The primary endpoint measurements are reported as areas under the curves (AUC) within the predefined range of acceptable respiratory parameters. Between-group differences in continuous variables are analysed using independent t-test or Mann-Whitney U test. Between-group differences in categorical variables are analysed using chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Decision made by treating physicians to intubate and mechanically ventilate

Exclusion Criteria:

1. Suspected or confirmed pregnancy.
2. Known right ventricular heart failure upon assessment for recruitment.
3. Severe metabolic acidosis upon intubation (pH <7.2 or bicarbonate <12 mmol/L)
4. Circulatory shock requiring noradrenaline more than 0.5 mcg/kg/min upon assessment for recruitment.
5. Severe or acute life-threatening asthma.
6. Patients with chest wall deformities that would affect ventilation (e.g. severe kyphoscoliosis, diaphragmatic hernia, flail chest, trauma, pectus excavatum or carinatum, ankylosing spondylitis
7. Patients with previous lobectomy or pneumonectomy.
8. Patients with pneumothorax or other condition that requires chest drainage tube.
9. Patients with body mass index > 40 kg/m2.
10. Manufacturer's contraindications:

    * Difference in oxygen saturation between pulse oximetry (SpO2) and arterial sample (SaO2) of more than 5% (due to unreliable sensor).
    * Difference in carbon dioxide level between end-tidal sensor (ETCO2) and arterial sample (PaCO2) of more than 5 mm Hg (due to unreliable sensor).
    * Known pneumothorax and bronchopulmonary fistula upon assessment for recruitment.
11. Participation in another interventional trial.
12. Do-not-attempt-resuscitation (DNAR) order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of ventilation within a predefined range of acceptable respiratory parameters | Every 30 seconds for 240 minutes
  Duration of ventilation (in minutes) within predefined acceptable tidal volume (TV), plateau pressure, EtCO2 and SpO2

SECONDARY OUTCOMES:
Manual adjustments of ventilator settings | Any time the manual adjustment is performed throughout the 4-hour study period
  Frequency of manual adjustments of ventilator settings and the parameters requiring adjustments
Physiological data - blood pressure | Mean hourly for 4 hours
  Patient's blood pressure in mmHg
Physiological data - respiratory rate | Mean hourly for 4 hours
  Patient's respiratory rate in breaths per minute
Physiological data - heart rate | Mean hourly for 4 hours
  Patient's heart rate in beats per minute
Biochemical data - pH | Upon intubation, at 1-hour, 2-hour, 3-hour and 4-hour
  Arterial pH levels
Biochemical data - CO2 and O2 | Upon intubation, at 1-hour, 2-hour, 3-hour and 4-hour
  Arterial partial pressure of carbon dioxide and oxygen in mmHg
Biochemical data - bicarbonate | Upon intubation, at 1-hour, 2-hour, 3-hour and 4-hour
  Arterial bicarbonate levels in mmol/L
Patient outcome - mechanical ventilation | Assessed from time of intubation to time of successful extubation or death from any cause, whichever came first, assessed up to 28 days
  Duration of mechanical ventilation
Patient outcome - LOS ED | Assessed from time of triage to time patient leaves ED or death, whichever comes first, up to 7 days
  Length of stay in emergency department
Patient outcome - LOS ICU | Assessed from time of admission into the ICU to time of transfer to general ward or death, whichever comes first up to 28 days
  Length of intensive care unit stay
Patient outcome - LOS hospital | Assessed from time of triage in ED to time of discharge or in-hospital death, whichever comes first up to 28 days
  Length of hospital stay
Mortality rate | At 14 and 28 days after recruitment
  Number and percentage of deaths
Number of patients developing ARDS and pneumothorax | At anytime within the 4-hour intervention or upon discharge or diagnosis of complications
  Development of complications (pneumothorax, ARDS) during study and throughout admission
Ventilator data - airway pressures | Every 30 seconds for 240 minutes
  Ventilator parameters: mean and peak airway pressures in cmH20
Ventilator data - FiO2 | Every 30 seconds for 240 minutes
  Ventilator parameters: fraction of inspired oxygen (FiO2)

CONTACTS AND LOCATIONS:
Overall Officials: Khadijah Poh, MMed, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: No
Individual participant data for this study will not be made publicly available. However, summary results and study outcomes will be transparently reported in the form of aggregated data and CSV files. This approach ensures that key findings are accessible while respecting participant confidentiality.

REFERENCES:
- [Background] Lellouche F, Bouchard PA, Simard S, L'Her E, Wysocki M. Evaluation of fully automated ventilation: a randomized controlled study in post-cardiac surgery patients. Intensive Care Med. 2013 Mar;39(3):463-71. doi: 10.1007/s00134-012-2799-2. Epub 2013 Jan 22. PMID 23338569
- [Background] Savioli G, Ceresa IF, Gri N, Bavestrello Piccini G, Longhitano Y, Zanza C, Piccioni A, Esposito C, Ricevuti G, Bressan MA. Emergency Department Overcrowding: Understanding the Factors to Find Corresponding Solutions. J Pers Med. 2022 Feb 14;12(2):279. doi: 10.3390/jpm12020279. PMID 35207769
- [Background] Angotti LB, Richards JB, Fisher DF, Sankoff JD, Seigel TA, Al Ashry HS, Wilcox SR. Duration of Mechanical Ventilation in the Emergency Department. West J Emerg Med. 2017 Aug;18(5):972-979. doi: 10.5811/westjem.2017.5.34099. Epub 2017 Jul 11. PMID 28874952
- [Background] Arnal JM, Garnero A, Novonti D, Demory D, Ducros L, Berric A, Donati S, Corno G, Jaber S, Durand-Gasselin J. Feasibility study on full closed-loop control ventilation (IntelliVent-ASV) in ICU patients with acute respiratory failure: a prospective observational comparative study. Crit Care. 2013 Sep 11;17(5):R196. doi: 10.1186/cc12890. PMID 24025234
- [Background] Clavieras N, Wysocki M, Coisel Y, Galia F, Conseil M, Chanques G, Jung B, Arnal JM, Matecki S, Molinari N, Jaber S. Prospective randomized crossover study of a new closed-loop control system versus pressure support during weaning from mechanical ventilation. Anesthesiology. 2013 Sep;119(3):631-41. doi: 10.1097/ALN.0b013e3182952608. PMID 23619172
- [Background] Chelly J, Mazerand S, Jochmans S, Weyer CM, Pourcine F, Ellrodt O, Thieulot-Rolin N, Serbource-Goguel J, Sy O, Vong LVP, Monchi M. Automated vs. conventional ventilation in the ICU: a randomized controlled crossover trial comparing blood oxygen saturation during daily nursing procedures (I-NURSING). Crit Care. 2020 Jul 22;24(1):453. doi: 10.1186/s13054-020-03155-3. PMID 32698860